CLINICAL TRIAL: NCT02094144
Title: Health Benefits of a 6-month Brisk Walking Program in Sedentary Postmenopausal Women : a Randomized Controlled Trial
Brief Title: Health Benefits of a 6-month Brisk Walking Program in Sedentary Postmenopausal Women
Acronym: ACTIMARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8189
Record Dates: First submitted 2014-03-13; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Sedentary Lifestyle; Postmenopausal Women
Keywords: Sedentary; Physical activity; Brisk walking; Postmenopausal women; Body composition; Balance; Muscle strength; Depression, bone density; Nutrition; Biological effects
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise group (brisk walking program) (Other): The intervention is named brisk walking program. It consists on achieve 40 minutes of brisk walking 3d/wk for 6 months (two supervised sessions and one session performed one their own per week with a detailed program). The intensity of the program is adapted to the heart rate work and gradually increases over the 6-month program
  Interventions: Other: Brisk walking program
- control group (physical activity habits) (Other): The Intervention consists on maintain the lifestyle and especially their physical activity habits during 6 months
  Interventions: Other: physical activity habit

INTERVENTIONS:
Other: Brisk walking program — The intervention consists on achieve 40 minutes of brisk walking 3d/wk for 6 months (two supervised sessions and one session performed one their own per week with a detailed program). The intensity of the program is adapted to the heart rate work and gradually increases over the 6-month program
  Arms: exercise group (brisk walking program)
Other: physical activity habit — The Intervention consists on maintain the lifestyle and especially their physical activity habits during 6 months
  Arms: control group (physical activity habits)

SUMMARY:
Community-dwelling women aged 55 or over are recruited at public meetings aimed at promoting physical activity in postmenopausal women. Women are eligible and enrolled in the study if they have no significant disease affecting lower limb function and if they have a sedentary lifestyle. All study participants provide written informed consent to participate to the study.

Women are then randomized either to the control group (women have to maintain their lifestyle) or to the exercise group : 40 minutes of brisk walking 3d/wk for 6 months (two supervised sessions and one session performed one their own per week with a detailed program). The intensity of the program is adapted to the heart rate work and gradually increases over the 6-month program. The objective of the study is to determine the health benefits of brisk on walking ability, diet, muscle strength, balance, blood pressure, bone density, body weight, lean and fat mass, depression symptoms, behavioral, emotional responses, sleep quality, and biological indicators of health.

DETAILED DESCRIPTION:
Community-dwelling women aged 55 or over are recruited at public meetings aimed at promoting physical activity in postmenopausal women.

Women are eligible and enrolled in the study if they meet the following criteria : (i) not diagnosed with any of the following conditions: rheumatoid arthritis, osteoarthritis, ischemic heart disease, previous joint replacement surgery or cerebrovascular disease affecting lower limb function, malignant tumors, (ii) without pain and medication known to alter physical performance (e.g., corticosteroids, estrogens, statins, or anti-estrogen drugs). To recruit a sample of asymptomatic sedentary postmenopausal women, women with a score value above 9.4 at the Physical Activity Questionnaire for the Elderly (PAQE) (Serres, Gautier, Varray, & Préfaut, 1998) and a 5-minute walking distance (6MWD) greater than105% of the predicted 6MWD based on Troosters' reference equation are excluded. The Troosters' reference equation is:

Before entering the study, women are asked to provide a medical certificate of no contraindication to performing the 6MWD.

Women are then randomized either to the control group (women are asked to maintain their lifestyle, and especially their physical activity habits) or to the exercise group.

The exercise intervention consists in 40 minutes of brisk walking 3d/wk for 6 months. During the 6-month program, subjects are required to attend 2 outdoor supervised sessions per week, and to exercise 1d/wk on their own, with a detailed and tailored program. The intensity of walking is adapted by skilled exercise trainers to individual physical capability of each subject. Considering that the theoretical maximum heart rate (HR) of the subject is 208-0.7 * age (Tanaka, Monahan, & Seals, 2001), the training starts at 40% of HR work (difference between maximum HR and HR at rest). Training intensity is gradually increased to finally reaching 75% of the HR work. Participants wear a heart rate monitor (Polar Elctro Inc, Woodbury, NY) during each of the 3 weekly sessions and the content of each session is collected in a notebook (meters walked, duration of the brisk walking exercise, HR, adherence to the program).

This study is approved by the Committee for Protection of Human Subjects (CPP Sud-Méditerranée III, Number: 2008.07.04). All study participants provide a written informed consent to participating to the study.

The objectives of the study are to determine the health benefits of the intervention program in comparison to the control group in several domains.

Mesurements at baseline and at the end of the study comprise:

* Body composition (bone density, body lean and fat mass by dual-energy X-ray absorptiometry (DXA) (Hologic QDR-1500 device, Hologic, Waltham, MA, USA);
* The subjects are weighed on an electronic scale to the nearest 0.1 kg, and their height is measured to the nearest 0.1 cm to calculate the body mass index (BMI)(kg/m²).
* Endurance training performance is estimated by the distance walked during the 6-minute walk test (6MWT). The 6MWT is performed according to the American Thoracic Society (2002) guidelines in an indoor corridor (ATS, 2002).
* Maximum grip strength and isometric maximum knee extension strength are measured after a warm-up session, as previously described (Blain et al., 2010).
* The Diet over the previous 7 days using the questionnaire used in the SUVIMAX study
* Sleep quality
* Depression score : French version of the Beck Depression Inventory (BDI) (Beck, Steer, & Carbin, 1988; Cathébras, Mosnier, Lévy, Bouchou, & Rousset, 1994). The BDI contains cognitive (e.g., pessimism, worthlessness) and physical (e.g., fatigue and loss of energy) subscales. The BDI has been shown to be sensitive to exercise-induced changes in healthy adults (Stein & Motta, 1992).
* Baseline physical activity, covering household activities, sports, and leisure activities is assessed using PAQE (Voorrips, Ravelli, Dongelmans, Deurenberg, & Van Staveren, 1991). The activities of walking outside, bicycling, and doing heavy housework are summed to a physical activity score (range, 0-3). Respondents not participating in any activity are given zero points, whereas three points corresponds to participation in all three activities.
* Subjective health status is assessed with the following item: In comparison to people with the same age, you consider your health as better (1), equal (2), worst (3) ?.
* The Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that assesses the fear of (re)injury due to movement (Swinkels-Meewisse, Swinkels, Verbeek, Vlaeyen, & Oostendorp, 2003). Women are asked to make ratings of their degree of agreement with each of the 17 statements. Ratings are summed to yield a total score where higher values reflect greater fear of (re)injury (French, France, Vigneau, French, & Evans, 2007).
* Balance is assessed using a force platform (Medicapteurs France SAS) with two conditions tested, eyes open (EO) and eyes closed (EC), lasting 51.2 seconds each and separated by a 30-second rest period. The COP trajectories in antero-posterior (AP) and medio-lateral (ML) directions are sampled at 40 Hz, leading time series with length of 2048.

Traditional stabilometric measures : the AP and ML standard deviations (SDx and SDy, mm), the effective COP path length (mm), and the area of the 90% confidence ellipse enclosing the COP (mm²).

Complexity measures of postural sway : The complexity of postural sway is quantified by means of three measures : Percentage of determinism of recurrence quantification analysis (DETRQA) , Sample entropy (SampEn), Complexity index of multiscale entropy (CIMSE)

* The adherence rate to the brisk walking program is calculated based on the data recorded in the notebooks (number of supervised and self-reported home based walking sessions performed/72 sessions of the program).
* Individual content of the training (meters walked measured with a podometer; total duration of the walking exercises, mean HR, etc…).
* Fasted morning blood samples are collected at baseline and at the end of the study and aliquots are frozen at -80 °C until analysis.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women aged 55 or older
* women were asked to provide a medical certificate of no contraindication to performing the 6MWD.

Exclusion Criteria:

* rheumatoid arthritis, osteoarthritis, ischemic heart disease, previous joint replacement surgery or cerebrovascular disease affecting lower limb function, malignant tumors, any pain or medication known to alter physical performance (e.g., corticosteroids, estrogens, statins, or anti-estrogen drugs)
* score value above 9.4 at the Physical Activity Questionnaire for the Elderly
* a 6MWD greater than 105% of the predicted 6MWD based on Troosters' reference equation

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
6 minute-walking distance (6MDWS) | 6 months
  6MWD was performed following ATS guidelines

SECONDARY OUTCOMES:
Effect of the brisk walking program on body composition | 6 months
  Assesment of lean body mass and fat body mass
Effect of the brisk walking program on depression symptoms | 6 months
  assessment with specific scale
Effect of the brisk walking program on muscle strength | 6 months
Effect of the brisk walking program on biological parameters | 6 months
  measure of PTH, calcitriol (1,25 OHD)
Effect of the brisk walking program on sleep quality | 6 months
  Assessment with specific scale

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Blain, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France